CLINICAL TRIAL: NCT05708989
Title: Caudal vs. Pudendal Block for Early Postoperative Pain Control in a Pediatric Population Undergoing Lower Genitourinary Surgery
Brief Title: Caudal vs. Pudendal Block in Peds GU
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20220033
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Hypospadias; Penile Torsion; Chordee; Phimosis
Keywords: caudal block; pudendal block; regional anesthesia
MeSH Terms: conditions — Hypospadias; Phimosis | interventions — Injections; Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caudal Block (Active Comparator): Patients will receive a caudal block prior to surgery.
  Interventions: Procedure: Caudal Block; Drug: Injectable 1 ml/kg of 0.25% ropivacaine with 1mcg/kg dexmedetomidine
- Pudendal Block (Experimental): Patients will receive a pudendal block prior to surgery.
  Interventions: Procedure: Ultrasound-guided Pudendal Block; Drug: Injection of 0.5 ml/kg per side of injectable 0.2-0.3% ropivacaine with 0.5 mcg/kg dexmetomedine.

INTERVENTIONS:
Procedure: Caudal Block — Injectable 1 ml/kg of 0.25% ropivacaine with 1mcg/kg dexmedetomidine into caudal spinal space. First attempt will be landmark-guided into the caudal spine region. Subsequent attempt(s) may be done using ultrasound.
  Arms: Caudal Block
Procedure: Ultrasound-guided Pudendal Block — Injection of 0.5 ml/kg per side of injectable 0.2-0.3% ropivacaine with 0.5 mcg/kg dexmetomedine. Ultrasound-guided injection into each pudendal nerve region through skin of buttocks.
  Arms: Pudendal Block
Drug: Injectable 1 ml/kg of 0.25% ropivacaine with 1mcg/kg dexmedetomidine — Injectable 1 ml/kg of 0.25% ropivacaine with 1mcg/kg dexmedetomidine into caudal spinal space. First attempt will be landmark-guided into the caudal spine region. Subsequent attempt(s) may be done using ultrasound.
  Arms: Caudal Block
Drug: Injection of 0.5 ml/kg per side of injectable 0.2-0.3% ropivacaine with 0.5 mcg/kg dexmetomedine. — Injection of 0.5 ml/kg per side of injectable 0.2-0.3% ropivacaine with 0.5 mcg/kg dexmetomedine. Ultrasound-guided injection into each pudendal nerve region through skin of buttocks.
  Arms: Pudendal Block

SUMMARY:
This study will compare two techniques to minimize pain during and after penile surgery in children undergoing certain urologic surgeries. These two approaches include the caudal nerve block and the pudendal nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing penile genitourinary surgery
* ASA class 1-3

Exclusion Criteria:

* Female patients
* Male children <6 months or >/= 3 years of age
* ASA class >3
* Surgery at satellite location (non-Prentiss)
* Concurrent non-lower GU tract surgery
* Sacrospinal abnormality
* History of chronic pain requiring opioid analgesics
* Inability to tolerate and receive acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), alpha-2 agonists, or local anesthetics
* History of malignant hyperthermia
* History of coagulopathy

Ages: 6 Months to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Rescue Narcotic Administration | During post-operative in-hospital recovery, approximately 1 hour
  Dose (mg) of postoperative rescue opioid

SECONDARY OUTCOMES:
Non-Narcotic Rescue Administration at 24 hours | During first day after surgery, approximately 24 hours
  Dose (mg) of non-narcotic rescue medication
Non-Narcotic Rescue Administration at 48 hours | During second day after surgery, approximately 48 hours
  Dose (mg) of non-narcotic rescue medication
Non-Narcotic Rescue Administration at 72 hours | During third day after surgery, approximately 72 hours
  Dose (mg) of non-narcotic rescue medication
Number of participants with at least one adverse event (AE) as measured by patient report | End of study, up to 3 months
  Adverse events will include any AE related to study procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jessica H Hannick, MD, MSc, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- UH Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wren AA, Ross AC, D'Souza G, Almgren C, Feinstein A, Marshall A, Golianu B. Multidisciplinary Pain Management for Pediatric Patients with Acute and Chronic Pain: A Foundational Treatment Approach When Prescribing Opioids. Children (Basel). 2019 Feb 21;6(2):33. doi: 10.3390/children6020033. PMID 30795645
- [Background] Vargas A, Sawardekar A, Suresh S. Updates on pediatric regional anesthesia safety data. Curr Opin Anaesthesiol. 2019 Oct;32(5):649-652. doi: 10.1097/ACO.0000000000000768. PMID 31415045
- [Background] Wiegele M, Marhofer P, Lonnqvist PA. Caudal epidural blocks in paediatric patients: a review and practical considerations. Br J Anaesth. 2019 Apr;122(4):509-517. doi: 10.1016/j.bja.2018.11.030. Epub 2019 Feb 1. PMID 30857607
- [Background] Okoro C, Huang H, Cannon S, Low D, Liston DE, Richards MJ, Lendvay TS. The pudendal nerve block for ambulatory urology: What's old is new again. A quality improvement project. J Pediatr Urol. 2020 Oct;16(5):594.e1-594.e7. doi: 10.1016/j.jpurol.2020.07.025. Epub 2020 Jul 24. PMID 32819811
- [Background] Shah UJ, Nguyen D, Karuppiaah N, Martin J, Sehmbi H. Efficacy and safety of caudal dexmedetomidine in pediatric infra-umbilical surgery: a meta-analysis and trial-sequential analysis of randomized controlled trials. Reg Anesth Pain Med. 2021 May;46(5):422-432. doi: 10.1136/rapm-2020-102024. Epub 2021 Jan 15. PMID 33452203
- [Background] Gaudet-Ferrand I, De La Arena P, Bringuier S, Raux O, Hertz L, Kalfa N, Sola C, Dadure C. Ultrasound-guided pudendal nerve block in children: A new technique of ultrasound-guided transperineal approach. Paediatr Anaesth. 2018 Jan;28(1):53-58. doi: 10.1111/pan.13286. Epub 2017 Dec 5. PMID 29205687
- [Background] Kendigelen P, Tutuncu AC, Emre S, Altindas F, Kaya G. Pudendal Versus Caudal Block in Children Undergoing Hypospadias Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):610-5. doi: 10.1097/AAP.0000000000000447. PMID 27501015
- [Background] Naja ZM, Ziade FM, Kamel R, El-Kayali S, Daoud N, El-Rajab MA. The effectiveness of pudendal nerve block versus caudal block anesthesia for hypospadias in children. Anesth Analg. 2013 Dec;117(6):1401-7. doi: 10.1213/ANE.0b013e3182a8ee52. PMID 24257391